CLINICAL TRIAL: NCT04887363
Title: The Comparisons of Effects of Core Stability Exercise and Tai Chi on Core Muscle Performances, Core Stability and Balance in Community-living Elderly
Brief Title: The Comparisons of Effects of Core Stability Exercise and Tai Chi on Core Muscle Performances in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KMUH-IRB-20120427
Record Dates: First submitted 2021-03-22; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-02

CONDITIONS: Tai Ji
MeSH Terms: interventions — Aquatic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Core exercise group (Experimental): The healthy community-dwelling older adults (60-74 years old), who had not received any core stability or Tai Chi Chuan training within the previous 6 months, were recruited in this study. All the subjects were independent in basic daily living activities and able to move freely without any assistance.
  Interventions: Behavioral: Core exercise
- Tai Chi exercise group (Experimental): The healthy community-dwelling older adults (60-74 years old), who had not received any core stability or Tai Chi Chuan training within the previous 6 months, were recruited in this study. All the subjects were independent in basic daily living activities and able to move freely without any assistance.
  Interventions: Behavioral: Tai Chi exercise
- Young adults group (No Intervention): The healthy young adults who have not any neurological, musculoskeletal or rheumatic disease were recruited as a reference group. They would not receive any training program in the study.

INTERVENTIONS:
Behavioral: Core exercise — Participants will receive12-week, 60 minutes, 36-session exercise-based core stability training class. Participants need complete baseline assessments of muscle performance, and balance ability measures 1 week prior and 1 week and 12 weeks following the intervention. All subjects will receive two post-exercise measurements at 13th week and 25th week.
  Arms: Core exercise group
Behavioral: Tai Chi exercise — Participants will receive 12-week, 60 minutes, 36-session Tai Chi exercise training class. Participants need complete baseline assessments of muscle performance, and balance ability measures 1 week prior and 1 week and 12 weeks following the intervention. All subjects will receive two post-exercise measurements at 13th week and 25th week.
  Arms: Tai Chi exercise group

SUMMARY:
Core muscles and core stability has a key component in the postural control or balance. However, no clear evidence has been found for the positive relationship between core stability and postural control in the elderly, and the effects of core stabilizing training on postural control or balance in the elderly. The purposes of this project are to investigate the effects of core stability training program on muscle strength, muscle performance, and balance outcomes in elderly adults.

DETAILED DESCRIPTION:
In this pretest, posttest design study, elderly adults enrolled and assigned to the core exercise group or Tai Chi exercise group, the core exercise group received core exercise intervention comparing to Tai Chi exercise group participated Tai chi exercise program as a control group.

The young adults group were also enrolled for a reference group, not received any exercise intervention and just only received the measurements once.

Participants in the two elderly group will receive 12-week, 36-session exercise-based core stability training class. The each 60 minutes core exercise class focuses on exercise for improving strength, endurance of core muscles and trunk stability.

Participants need complete baseline assessments of muscle performance, and balance ability measures 1 week prior and 1 week and 12 weeks following the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Core exercise group and Tai Chi exercise group

   1. healthy community-dwelling older adults (60-74 years old)
   2. not received any core stability or Tai Chi Chuan training within the previous 6 months
   3. independent in basic daily living activities
   4. able to move freely without any assistance
2. Young adults group a. Their age should be ranged between 20 - 59 years

Exclusion Criteria:

All group

1. have a history of orthopedic surgery on spine or lower extremity
2. have any spine pathology (e.g., spondylolisthesis, disc herniation)
3. have a pain over back or lower limbs to affect the ability to perform activities of daily living
4. had a history of vestibular disease (e.g., Meniere' s disease)

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-06-03 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in strength of core muscle groups (trunk) at 12-week | The assessments will be conducted 1 and 12 weeks following the intervention
  Using a custom-made isometric dynamometer to measure the strength of trunk flexors, extensors and rotators
Changes in strength of core muscle groups (hip) at 12-week | The assessments will be conducted 1 and 12 weeks following the intervention
  Using a hand-held dynamometer to measure the hip muscle strength
Changes in endurance of core muscle groups at 12-week | The assessments will be conducted 1 and 12 weeks following the intervention
  Using the Stabilizer Pressure Biofeedback Unit (PBU) during the leg-loading test to measure the endurance of lumbo-pelvic stability
Changes in flexibility of the lower back and hamstring muscles at 12-week | The assessments will be conducted 1 and 12 weeks following the intervention
  Using the sit and reach test to measure the flexibility of the lower back and hamstring muscles
Changes in ability of the dynamic balance at 12-week | The assessments will be conducted 1 and 12 weeks following the intervention
  Using the Dual-tasking 3m Timed up and go (3m-TUG) to measure dynamic balance and the fall risk. Mean time to perform 3m-TUG is 11.56 seconds
Changes in assessment of postural control at 12-week | The assessments will be conducted 1 and 12 weeks following the intervention
  Using a force plate to collect the center of pressure (COP) displacement
Changes in muscle activity of selected core muscles during performing arm-raising tasks at 12-week | The assessments will be conducted 1 and 12 weeks following the intervention
  Using a surface electromyography to record the muscle activity of abdominal and trunk muscles during performing arms-raising tasks with hand-holding 1.5-2 kg
Changes in assessment of postural control during performing arm-raising tasks at 12-week | The assessments will be conducted 1 and 12 weeks following the intervention
  Using a force plate to collect the center of pressure (COP) displacement during performing arms-raising tasks with hand-holding 1.5-2 kg

CONTACTS AND LOCATIONS:
Overall Officials: Li-Jiun Liaw, Study Director — Kaohsiung Medical University Department of Physical Therapy Associate Professor

IPD SHARING:
Plan to Share IPD: No
Currently in the submission stage ,and then share with other researchers after publication